CLINICAL TRIAL: NCT06662110
Title: A Prospective Cohort Study on Serum Immune Protein Signature for Predicting Neoadjuvant Therapy Efficacy in Advanced Gastric Cancer
Brief Title: IMmune Proteomics to Predict NeoAdjuvant Chemotherapy and ImmunoTherapy Response in Gastric Cancer
Acronym: IMPACT-GC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IMPACT-GC
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 1. peripheral blood of patients
  2. tumor tissue specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- neoadjuvant chemotherapy cohort: Resectable gastric cancer patients who received neoadjuvant chemotherapy, with the SOX regimen as the representative treatment plan, in accordance with standard clinical practice.
  Interventions: Diagnostic Test: PSRscore
- neoadjuvant chemotherapy plus immunotherapy cohort: Resectable gastric cancer patients who received neoadjuvant chemotherapy plus immunotherapy in accordance with standard clinical practice.
  Interventions: Diagnostic Test: PSRscore

INTERVENTIONS:
Diagnostic Test: PSRscore — PSRscore calculated based on baseline serum immune proteomics

SUMMARY:
The overall efficacy of neoadjuvant treatment for advanced gastric cancer is limited due to significant heterogeneity in patient responses. While neoadjuvant therapy offers hope for improved clinical outcomes, the key challenge is accurately predicting individual treatment responses. Identifying reliable biomarkers to guide treatment decisions is therefore critical. Immune factors are pivotal in the efficacy of gastric cancer treatment, but most research has predominantly focused on the tumor immune microenvironment. This study aims to validate the predictive value of systemic immune markers in predicting neoadjuvant treatment responses in advanced gastric cancer.

Building on our previous research, where we established a retrospective cohort of patients with advanced gastric cancer undergoing preoperative chemotherapy, we employed a novel serum proteomics platform based on proximity extension assays (PEA) to measure key immune protein levels in patient serum. This led to the development of the PSRscore system, a serum immune protein score that effectively predicted tumor regression after preoperative chemotherapy (published in Cell Reports Medicine, doi: 10.1016/j.xcrm.2023.100931).

In this prospective cohort study, we will enroll 166 patients with resectable advanced gastric cancer undergoing neoadjuvant chemotherapy. Baseline serum samples will be collected prior to treatment, and the PSRscore will be used to predict tumor regression. Pathological evaluation post-chemotherapy will confirm tumor response, helping to further validate and refine the PSRscore system. Additionally, an exploratory cohort of 40 patients receiving combined neoadjuvant chemotherapy and immunotherapy will be included to evaluate the correlation between PSRscore and clinical benefit from immunotherapy.

This research is expected to lead to the development of a predictive diagnostic kit based on the PSRscore for advanced gastric cancer patients undergoing neoadjuvant therapy, with the ultimate goal of improving clinical decision-making and enhancing treatment outcomes for gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria

1. Males or females aged 18 to 75 years;
2. Newly diagnosed histologically confirmed gastric adenocarcinoma;
3. Lesion located in the stomach or gastroesophageal junction as assessed by endoscopic ultrasound and enhanced CT, with clinical staging of T3-4NxM0 (based on the 8th edition of AJCC TNM classification);
4. Determined suitable for neoadjuvant chemotherapy or neoadjuvant chemotherapy combined with immunotherapy after multidisciplinary consultation, with potential for curative resection post-treatment. The chemotherapy regimen is restricted to fluoropyrimidine and platinum-based systemic chemotherapy; the immunotherapy regimen is restricted to immune checkpoint inhibitors.

Exclusion Criteria

1. Prior receipt of any anti-tumor therapy for current gastric cancer or receipt of anti-tumor drugs for other conditions within the past 4 weeks;
2. Presence of another malignancy or multiple primary tumors;
3. Serious comorbidities with a life expectancy of less than 5 years;
4. Severe chronic or active infections requiring systemic anti-infective therapy;
5. Blood transfusion within the past week;
6. Receipt of corticosteroid or immunosuppressive therapy within the past 2 weeks;
7. Administration of a live vaccine within the past 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable gastric cancer patients who received neoadjuvant treatment followed by gastrectomy with D2 lymphadenectomy at Zhongshan Hospital, Fudan University
Sampling Method: Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
the sensitivity and specificity of PSRscore in predicting tumor regression after neoadjuvant therapy in patients with advanced gastric cancer | From enrollment to the end of the pathological examination of all resected tumor samples, an average of 2 years

SECONDARY OUTCOMES:
the sensitivity and specificity of PSRscore in predicting objective response after neoadjuvant treatment in patients with advanced gastric cancer | From enrollment to the end of all the neo-adjuvant treatment, an average of 2 years
the sensitivity and specificity of PSRscore in predicting progression-free survival (PFS) after neoadjuvant treatment in patients with advanced gastric cancer | though study completion, an average of 5 years
the sensitivity and specificity of PSRscore in predicting overall survival (OS) after neoadjuvant treatment in patients with advanced gastric cancer | though study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, Principal Investigator — Fudan University; Zhaoqing Tang, Principal Investigator — Fudan University; Yuan Gu, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Xuhui District, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang Z, Gu Y, Shi Z, Min L, Zhang Z, Zhou P, Luo R, Wang Y, Cui Y, Sun Y, Wang X. Multiplex immune profiling reveals the role of serum immune proteomics in predicting response to preoperative chemotherapy of gastric cancer. Cell Rep Med. 2023 Feb 21;4(2):100931. doi: 10.1016/j.xcrm.2023.100931. Epub 2023 Jan 31. PMID 36724786